CLINICAL TRIAL: NCT05657028
Title: Intravenous Dexmedetomidine Versus Intravenous Lidocaine in Attenuating Airway Reflexes During Recovery of Thyroidectomy Patients
Brief Title: Dexmedetomidine Versus Lidocaine in Attenuating Airway Reflexes During Recovery of Thyroidectomy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: attenuating airway reflexes
Record Dates: First submitted 2022-11-08; First posted 2022-12-20 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia; Airway Complication of Anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Dexmedetomidine) (Experimental): In the Dexmedetomidine group, patients will be given IV bolus infusion of dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- Group L (Lidocaine) (Experimental): In the Lidocaine group, the patients will be given an IV bolus infusion of lidocaine
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Dexmedetomidine — -In the Dexmedetomidine group, patients will be given IV bolus infusion of dexmedetomidine 0.5 μg/kg over 10 min before induction of anesthesia, followed by a continuous IV infusion of dexmedetomidine 0.4 μg/kg/hour until 30 min before the end of surgery.
  Arms: Group D (Dexmedetomidine)
Drug: Lidocaine IV — In the Lidocaine group, the patients will be given an IV bolus infusion of lidocaine (2%)1.5mg/kg over 10 min before induction of anesthesia, followed by a continuous IV infusion of lidocaine 1.5 mg/kg /hour until 30 min before the end of surgery.
  Arms: Group L (Lidocaine)

SUMMARY:
It is widely believed that most of the patients experience a cough upon emergence from general anesthesia, due to many causes including the presence of an endotracheal tube, uncleared secretions and anesthetic gas. Cough during tracheal extubation may lead to several complications, such as hypertension, tachycardia and postoperative bleeding.

In this study the investigators are going to compare the effectiveness of intravenous Dexmedetomidine and intravenous lidocaine in attenuating the air way reflexes and coughing during recovery of thyroidectomy patients.

DETAILED DESCRIPTION:
Intubation and extubation process are associated with cardiovascular and various airway responses leading to tachycardia, hypertension, arrhythmia, myocardial ischemia, cough induction, bronchospasm, increased bleeding, increased intracranial and intraocular pressure. Causes possibly include the presence of an endotracheal tube, uncleared secretions, and anesthetic gas.

Furthermore, postoperative bleeding in thyroid surgery is still significant and is often associated with severe complications including cervical hematoma, reoperation and cardiac arrest.

Extubation under deep anesthesia decreases cardiovascular stimulation and reduces the incidence of coughing and straining on the tube. Intratracheal local anesthetic instillation, I.V lidocaine, short acting opioids such as fentanyl and remifentanil, esmolol, labetalol, diltiazem and verapamil have been used to attenuate these hemodynamic and respiratory responses during extubation in the past but with certain limitations.

Also "no stimulation" extubation technique avoids extubation under light anesthesia and ensures extubation only when consciousness is returned. It requires absolutely no stimulation during emergence and performing extubation only when the patient wakes up spontaneously and opens his eyes.

Recently dexmedetomidine, a potent α2-adrenoreceptor agonist has been used to facilitate extubation in surgical intensive care unit, but its role in the attenuation of hemodynamic and airway reflexes during extubation in general anesthesia is still under study.

In this study the investigators are going to compare the effects of intravenous lidocaine and dexmedetomidine in inhibiting cough reflex during the recovery period after thyroid surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective thyroidectomy surgery.
* Age: patients between 18-and 65-years old from both sexes.
* Classified as either American Society of Anesthesiologists (ASA) class I or II.

Exclusion Criteria:

* Refusal of procedure or participation in the study.
* Patients suffering from asthma, chronic cough, preoperative upper respiratory infection symptoms.
* Current smoker.
* Medication involving angiotensin-converting-enzyme inhibitors (ACE-I).
* Classified as either American Society of Anesthesiologists (ASA) class III or IV.
* Sinus Bradycardia (<60/min) or history of any type of heart block or Beta-Blockers medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
compare effectiveness of Dexmedetomidine and intravenous lidocaine in attenuating cough reflex during the tracheal extubation period after thyroid surgery | 5 minutes from extubation
  the investigators use the following cough score where 0 = no cough, 1 = minimal (single) cough, 2 = moderate (≤5 seconds) cough and 3 = severe (>5 seconds) cough to reflect the degree of attenuation of air way reflexes for each group

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hu S, Li Y, Wang S, Xu S, Ju X, Ma L. Effects of intravenous infusion of lidocaine and dexmedetomidine on inhibiting cough during the tracheal extubation period after thyroid surgery. BMC Anesthesiol. 2019 May 4;19(1):66. doi: 10.1186/s12871-019-0739-1. PMID 31054568